CLINICAL TRIAL: NCT06317181
Title: Acquisition and Frequency Spectroscopic Evaluation of Broadband Clinical Ultrasound Raw Data for Liver Cirrhosis and Focal Pathologies Using Neural Networks for Tissue and Pathology Differentiation
Brief Title: Assessment of Liver Diseases Using a Deep-Learning Approach Based on Ultrasound RF-Data
Acronym: LivSPECTRUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Dresden (Other); University of Leipzig (Other)
Responsible Party: Principal Investigator, Moritz Herzog, Principal Investigator, Technische Universität Dresden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DifLivSPECTRUS
Record Dates: First submitted 2024-03-01; First posted 2024-03-19 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Artificial Intelligence; Ultrasonography; Elasticity Imaging Techniques; Liver Diseases; Metastasis to Liver
Keywords: Quantitative Ultrasound; Radiofrequency Data
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: Data is collected in a defined group of patients (all patients listed for elastography or for ultrasonic investigation due to a focal lesion in participating departments). Afterwards performances of algorithms are compared based on this group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elastography (Experimental): Collection of ultrasound data and elastography data from patients who were clinically planned for elastography
  Interventions: Device: Collection of elastography data
- Focal lesion (Experimental): Collection of ultrasound data of the suspected lesion and a definitive diagnosis based on either normal ultrasound investigation or if not sufficient additional investigations like CEUS, Biopsy, MRI or CT. This further investigation should be in accordance to normal clinical routine of the centers to differentiate focal lesions.
  Interventions: Device: Collection of ultrasonic raw data

INTERVENTIONS:
Device: Collection of elastography data — patients who are scheduled for an elastography for clinical reasons usually receive an ultrasound scan in which the b-mode images of the liver tissue are collected. In this study additional radiofrequency data is collected through a software access.
  Arms: Elastography
Device: Collection of ultrasonic raw data — Patients who are transferred to the ultrasound departement due to suspicious focal lesions receive an ultrasonic investigation including the acquisition of raw data and extracting a definitive diagnose from the following clinical routine investigation, depending on the standards of the participating center
  Arms: Focal lesion

SUMMARY:
The goal of this clinical trial is to test the performance of neuronal networks trained on ultrasonic raw Data (=radiofrequency data) for the assessment of liver diseases in patients undergoing a clinical ultrasound examination. The general feasibility is currently evaluated in a retrospective cohort.

The main questions the study aims to answer are:

* Can a neuronal network trained on RF Data perform equally good as elastography in the assessment of diffuse liver diseases?
* Can a neuronal network trained on RF Data perform better than a neuronal network trained on b-mode images in the assessment of diffuse liver diseases?
* Can a neuronal network trained on RF Data distinguish focal pathologies in the liver from healthy tissue?

To answer these questions participants with a clinically indicated fibroscan will undergo:

* a clinical elastography in Case ob suspected diffuse liver disease
* a reliable ground truth (if normal ultrasound is not sufficient e.g. contrast enhanced ultrasound, biopsy, MRI or CT) in case of focal liver diseases, depending on the standard routine of the participating center
* a clinical ultrasound examination during which b-mode images and the corresponding RF-Data sets are captured

ELIGIBILITY:
Inclusion Criteria:

* scheduled for an ultrasound investigation by an independent physician
* signed declaration of consent

Exclusion Criteria:

* smaller interventions in the same liver during the last 2 Week (for example liver biopsy)
* contrast enhanced ultrasound less than a day ago
* major intervention at the liver (for example partial resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Performance analysis of the trained model | After study completion, estimated 1 year
  Analysis of the concordance of a Deep Learning-based analysis of RF data with established clinical measures. In case of diffuse disease the stiffness of the tissue and in case of the focal lesions the underlying disease as diagnosed by the local physicians are the measures.
  Performance is evaluated by the area under the receiver operating characteristic curve and a correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Herzog, MD, Principal Investigator — University Hospital Dresden
Locations (4):
- Germany (4):
  - University Hospital, Dresden
  - Diakonissen Hospital Dresden, Dresden
  - University Hospital Halle (Saale), Halle
  - University Hospital Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: Yes
After the publication of data the anonymized IPD will be provided.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after finishing the study, data will be stored locally for at least 7 years
Access Criteria: contact the investigators via mail
URL: https://digitalhealth.tu-dresden.de/projects/hybridecho/spectrus/

REFERENCES:
- See also: Webpage of the project with updated information, participating partners and resulting publications — https://digitalhealth.tu-dresden.de/projects/hybridecho/spectrus/

DOCUMENTS (1):
  • Study Protocol (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT06317181/Prot_000.pdf